CLINICAL TRIAL: NCT02476032
Title: An Evaluation of the Efficacy of Oral-B New Product Sensi-Stop on Dentinal Hypersensitivity
Acronym: SSDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1503M65361
Record Dates: First submitted 2015-05-27; First posted 2015-06-19 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Tooth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prof applied oxalate (Experimental): Subjects will be randomized to either receive the Prof applied oxalate Crest Sensi-Stop strip (Procter & Gamble™). The oxalate strip contains 3% dipotassium oxalate desensitizing gel. The placebo strip is blank. The strips will be placed by a licensed dental professional and will be in place for 10 minutes. Subjects will be instructed to not rinse their mouth, drink, eat or brush their teeth for 30 minutes after completion of the treatment.
  Interventions: Device: Prof applied oxalate
- Self-applied oxalate (Active Comparator): Participants randomized to the Active Comparator Group will have the following intervention: Intervention: self-applied oxalate (Crest Sensi-Stop strip Procter & Gamble™), which contains 3% dipotassium oxalate desensitizing gel. The strip will be placed by the participant, following the manufacturer's directions. The strip will be left in place for 10 minutes. Subjects will be instructed to not rinse their mouth, drink, eat or brush their teeth for 30 minutes after completion of the treatment.
  Interventions: Device: Self applied oxalate
- Prof applied placebo (Sham Comparator): Subjects will be randomized to either receive the Prof applied placebo Crest Sensi-Stop strip (Procter & Gamble™). The oxalate strip contains 3% dipotassium oxalate desensitizing gel. The placebo strip is blank (sham). The strips will be placed by a licensed dental professional and will be in place for 10 minutes. Subjects will be instructed to not rinse their mouth, drink, eat or brush their teeth for 30 minutes after completion of the treatment.
  Interventions: Device: Prof applied placebo

INTERVENTIONS:
Device: Prof applied oxalate — Crest Sensi-Stop strips (Procter & Gamble™) with the active ingredient will be placed on the qualifying teeth by a dental professional.
  Arms: Prof applied oxalate
Device: Self applied oxalate — Subjects will apply the strips (Procter & Gamble™), that contain the active ingredient, by themselves following the manufacturer's instructions.
  Arms: Self-applied oxalate
Device: Prof applied placebo — Crest Sensi-Stop strips (Procter & Gamble™) without the active ingredient will be placed on the qualifying teeth by a dental professional.
  Arms: Prof applied placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of Sensi-StopTM strips (Procter & Gamble™) on the relief of dentinal hypersensitivity. In other words, do Sensi-StopTM strips (Procter & Gamble™) reduce or eliminate cold sensitivity in teeth? In addition, the investigators will evaluate whether there is a difference in the Sensi-StopTM strip (Procter & Gamble™) effectiveness when the product is placed by a dental professional compared to self-placement by the person with sensitive teeth. This product is not experimental.

DETAILED DESCRIPTION:
There are two groups in this research study: 1) The Self Applied group, and 2) the Professionally Applied group.

Once it is determined that interested individuals qualify to participate in the study and have determined that they want to participate, the group that participants are in will be determined. The study has been designed to ensure that 66% of the study participants receives strips that contain the active ingredient and 33% of the subjects receive strips without the active ingredient. This means that there is a 1 out of 3 chance that participants will be assigned to receive the strip(s) without the active desensitizing ingredient. At the end of your 8-week participation, if it turns out that participants received the strips without the active ingredient, they will be offered a sample pack with two strips that contain the active desensitizing ingredient for them to use at home.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents in good general health with no allergies to commercial dental products and are currently not using any desensitizing agents.
* If participants are using desensitizing agent the participant must agree to not use any desensitizing agents in the 4 weeks leading up to the baseline data collection appointment and during the following 8 week length of the study.
* Patients with a history of having used Sensi-Stop Strips (Procter & Gamble™) in the past will not be eligible to participate because it will not be possible to maintain blindness to the treatment that they receive.
* Patients will also have at least the following baseline measurements:

  i. Schiff Air Scale = equal to or greater than 1

ii. Verbal Rating Scale = equal to or greater than 1

iii. Recession= 1mm or greater

Exclusion Criteria:

* Any dental pathology resulting in pain that could confound the study findings would render the patient ineligible: e.g. advanced dental decay, pulpitis, fractured teeth, fractured restorations, chipped teeth, cracked teeth, severe gingival inflammation, post-restorative sensitivity, marginal leakage, severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession.
* Also, if potential study subjects are not willing to agree to avoid the use of desensitizing and/or whitening products they will not be enrolled.
* Adults lacking in the ability to give consent will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Lenton, MA, CCRP, Principal Investigator — University of Minnesota
Locations (1):
- Oral Health Research Clinic at the School of Dentistry at the University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
At this time, we do not plan to share individual participant data. We are willing to share compiled data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Prof Applied Oxalate: Subjects will be randomized to receive the Prof applied oxalate Crest Sensi-Stop strip (Procter & Gamble™). The oxalate strip contains 3% dipotassium oxalate desensitizing gel. The strips will be placed by a licensed dental professional and will be in place for 10 minutes. Subjects will be instructed to not rinse their mouth, drink, eat or brush their teeth for 30 minutes after completion of the treatment.
  Professionally applied Crest Sensi-Stop strips (Procter & Gamble™): Crest Sensi-Stop strips (Procter & Gamble™) with the active ingredient will be placed on the qualifying teeth by a dental professional.
- Self-applied Oxalate: Participants randomized to the Active Comparator Group will have the following intervention: Intervention is the self-applied Crest Sensi-Stop strip (Procter & Gamble™), which contains 3% dipotassium oxalate desensitizing gel. The strip will be placed by the participant, following the manufacturer's directions. The strip will be left in place for 10 minutes. Subjects will be instructed to not rinse their mouth, drink, eat or brush their teeth for 30 minutes after completion of the treatment.
  Self applied Crest Sensi-Stop strips (Procter & Gamble™): Subjects will apply the strips (Procter & Gamble™), that contain the active ingredient, by themselves following the manufacturer's instructions.
- Prof Applied Placebo: Subjects will be randomized to receive the Prof applied placebo Crest Sensi-Stop strip (Procter & Gamble™). The placebo strip is blank (sham). The strips will be placed by a licensed dental professional and will be in place for 10 minutes. Subjects will be instructed to not rinse their mouth, drink, eat or brush their teeth for 30 minutes after completion of the treatment.
Period: Overall Study
Arm/Group | Prof Applied Oxalate | Self-applied Oxalate | Prof Applied Placebo
Started | 20 | 20 | 20
Completed | 20 | 19 | 19
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prof Applied Oxalate | Self-applied Oxalate | Prof Applied Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 19 | 58
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (16.1) | 47.3 (12.0) | 40.3 (15.4) | 43.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 15 | 44
  Male | 7 | 4 | 5 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  White | 17 | 17 | 14 | 48
  African American | 2 | 3 | 4 | 9
  Asian | 0 | 0 | 1 | 1
  Hispanic/Latino | 1 | 1 | 0 | 2
  Native American | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Schiff Air Scale [Mean (Standard Deviation); unit: units on a scale] — Schiff Air Scale 0-3 Measurement of Dentinal Hypersensitivity
  0 Tooth/Patient did not respond to the air stimulus
  1. Tooth/Patient responded to the air stimulus but did not request discontinuation of the stimulus
  2. Tooth/Patient responded to the air stimulus and request discontinuation or moved from the stimulus
  3. Tooth/Patient responded to the air stimulus, considered the stimulus painful, and requested discontinuation of the stimulus
  units on a scale | 1.4 (0.8) | 2.3 (0.8) | 2.0 (0.9) | 1.9 (0.83)
Verbal Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Verbal Rating Scale 0-10 Measurement of Participant's Perception of Pain
  0 = No pain 1-3 = Mild Pain 4-6 = Moderate Pain 7-10 = Severe Pain
  units on a scale | 4.3 (1.9) | 6.5 (1.8) | 5.8 (2.1) | 5.5 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Schiff Air Test: Mean Reduction in Sensitivity Between Groups
Description: An analysis of covariance model was used to compare mean reduction in sensitivity scores (SAS and VRS) between groups at each post-treatment time point. A linear mixed effect model with group, time and baseline score as fixed effects and a random subject effect was used to compare the sensitivity outcomes between groups across time. The effect of location was also examined using this model.
  Schiff Air Scale 0-3 Measurement of Dentinal Hypersensitivity
  0 Tooth/Patient did not respond to the air stimulus
  1. Tooth/Patient responded to the air stimulus but did not request discontinuation of the stimulus
  2. Tooth/Patient responded to the air stimulus and request discontinuation or moved from the stimulus
  3. Tooth/Patient responded to the air stimulus, considered the stimulus painful, and requested discontinuation of the stimulus
Time Frame: 30 Minutes Post, 4 Weeks Post, 8 Weeks Post Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Prof Applied Oxalate | Self-applied Oxalate | Prof Applied Placebo
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  30 Minutes Post | -0.66 (0.23) | -1.12 (0.23) | -0.52 (0.22)
  4 Weeks Post | -1.11 (0.26) | -0.86 (0.26) | -0.22 (0.24)
  8 Weeks Post | -1.24 (0.26) | -1.12 (0.26) | -0.78 (0.25)
Statistical Analysis 1: Comparison: Prof Applied Oxalate vs Self-applied Oxalate vs Prof Applied Placebo; Within group comparisons: t-tests comparing the mean change to 0 were utilized. P-values less than 0.05 were considered statistically significant. SAS V9.3 (SAS Institute Inc., Cary, NC) was used for analysis. The sample size of 20 participants per group was based on having 90% power to detect a one standard deviation difference between the DO-strip groups and the placebo group means using ANOVA with a 0.05 level of significance; Test type: Other; p = 0.05, t-test, 2 sided — P-values for pairwise group comparisons were adjusted for multiple comparisons using the Tukey method

2. Secondary Outcome: Verbal Rating Scale: Mean Reduction in Sensitivity Between Groups
Description: An analysis of covariance model was used to compare mean reduction in sensitivity scores (SAS and VRS) between groups at each post-treatment time point. A linear mixed effect model with group, time and baseline score as fixed effects and a random subject effect was used to compare the sensitivity outcomes between groups across time. The effect of location was also examined using this model.
  Verbal Rating Scale 0-10 Measurement of Participant's Perception of Pain
  0 = No pain 1-3 = Mild Pain 4-6 = Moderate Pain 7-10 = Severe Pain
Time Frame: 30 Minutes Post, 4 Weeks Post, 8 Weeks Post Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Prof Applied Oxalate | Self-applied Oxalate | Prof Applied Placebo
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  30 Minutes Post | -1.27 (0.42) | -1.85 (0.41) | -0.83 (0.39)
  4 Weeks Post | -2.22 (0.51) | -1.34 (0.52) | -0.20 (0.48)
  8 Weeks Post | -2.26 (0.52) | -1.66 (0.52) | -1.33 (0.50)
Statistical Analysis 1: Comparison: Prof Applied Oxalate vs Self-applied Oxalate vs Prof Applied Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.05, t-test, 2 sided — P-values for pairwise group comparisons were adjusted for multiple comparisons using the Tukey method

ADVERSE EVENTS:
Time Frame: Entire length of study
Arm/Group | Prof Applied Oxalate | Self-applied Oxalate | Prof Applied Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No